CLINICAL TRIAL: NCT06235255
Title: A Pilot Intervention Study to Promote Functional Health in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seton Hall University (Other)
Responsible Party: Principal Investigator, Phyllis Hansell, Dr. Phyllis Hansell, Professor, Graduate Nursing Department, College of Nursing, Seton Hall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID#2024-514
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Health Behavior
Keywords: Functional Health Women
MeSH Terms: conditions — Health Behavior | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Guided Imagery Intervention (Experimental): Participants randomly assigned to this group will be provided with a MP3 Player which will have three guided imagery programs. The Guided Imagery Programs include: 1.Relaxation and Wellness; 2. Immune System Imagery and 3. Healing Trauma. The study measures are completed upon entry and 21 days post entry into the study and include: PKPCT and 21 days post entry into the study and include: PKPCT and the SF-36v2.
  Interventions: Behavioral: Guided Imagery
- Cognitive Power Intervention (Experimental): The participant is randomly assigned to this group completes The Power as Knowing Participation in Change (PKPCT) to determine: 1. Freedom to Act Intentionally; 2. Involvement in creating change; 3.Freedom to act intestinally and 4. My involvement in creating change. The study measures are completed upon entry and 21 days post entry into the study and include: PKPCT and the SF-36v2.
  Interventions: Behavioral: Cognitive Power Intervention
- Combined Guided Imagery and Cognitive Power Intervention (Experimental): The participants are randomly assigned to this group completes The Power as Knowing Participation in Change (PKPCT) and the Guided Imagery Intervention as described above. The study measures are completed upon entry and 21 days after entry and include the PKPCT and the SF-36v2.
  Interventions: Behavioral: Combined Guided Imagery and Cognitive Power Intervention
- Control Group (No intervention) (No Intervention): The participants are randomly assigned to this group complete all study measures PKPCT and the SF-36v2 measures upon entry into the study and 21 days after entry.

INTERVENTIONS:
Behavioral: Guided Imagery — The participant will complete the Guided Imagery Intervention for 21 consecutive days.
  Arms: Guided Imagery Intervention
Behavioral: Cognitive Power Intervention — The investigator with the subject uses the power profile generated by the PKPCT to generate goals that will positively affect functional health.
  Arms: Cognitive Power Intervention
Behavioral: Combined Guided Imagery and Cognitive Power Intervention — This intervention is a combination of the Guided Imagery Intervention in tandem with the Cognitive Power Intervention
  Arms: Combined Guided Imagery and Cognitive Power Intervention

SUMMARY:
The goal of this randomized clinical trial aims to pilot test the effectiveness' of three health promotion interventions for the achievement of optimal functional health in women.. The study interventions include: a Cognitive Power Intervention; a Guided Imagery Intervention and a third intervention that combines the two interventions. The interventions are compared to each other and to a control group in women to improve functional health health status.

DETAILED DESCRIPTION:
This pilot intervention study is focused on testing three interventions aimed at the improvement of functional health status in women compared to a control group.function. Regardless of one's age or health status the functional health of a person can be supported and improved. Higher functional health can help to prevent chronic conditions while promoting increased functional health. Higher functional health levels in women can affect not only the person, but also the functional health of their family and friends future patients who may benefit from their role modeling.

A health promoting lifestyle specifically refers to self-directed behaviors that may mitigate adverse health behaviors. According to Pender al (2010) health promoting functional health behaviors consist of six dimensions of health and include: physical activity, nutrition, responsibility, interpersonal relations, spiritual growth and stress management. Despite numerous studies on functional health in women there are no clinical intervention trials testing interventions to improve the level of Functional Health (Park, S. et al (2016); Hong, S.H. (2013); and Yang, N.Y. et al (2019). Power as knowing Participation in Change is a theory that is derived from Rogers, Science of Unitary human Beings. Barrett's (2003) theory focuses on power as freedom to act intestinally which is in sharp contrast to power-as-control. Power-as-freedom comes from and is associated with participating knowingly in life changes (Barrett, 2010). The phases of the theory include Involvement; freedom freedom; choices and awareness (Barrett, 1984). The theory has been operationalized with valid and reliable instrumentation through the Participation in Change Tool (PKPCT).

The Cognitive Power intervention on Health Function uses the PKPCT to determine the subject's power profile to set attainable goals to act intentionally to create specific changes in one's life aimed at the improvement of their health function. Barrett's theory has been used in numerous research studies yet t date none are randomized clinical trials. In the proposed study the subjects power profile is used to effectively deploy their power to best enable the improvement of health function.

The second intervention which is Guided Imagery is a therapeutic technique that aids individuals in therapy to focus on mental images to invoke feelings of relaxation which is based upon the mind-body connection which is considered an important factor a person's overall health Giacobbi, PR (2017). Guided Imagery is considered as complementary and alternative therapy that has been widely used to impact the body as well as the mind. Guided imagery has been used to address pain management, high blood pressure, cancer and other chronic conditions (Zech.N.2017) The literature suggests there is a complementary association between Guided Imagery and Power as Knowing Participation in Change and the outcome of improved health function. This pilot study will help to identify the effects and direction of data which also will be used to further strengthen the future study protocols These data are intended as preliminary data to be included in a large-scale study on minority women with chronic health conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Speaks reads and writes English
2. Between the ages of 18-60

Exclusion Criteria:

1. Chronic Illnesses 2 Cognitive Impairment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy females between 18-60 years of age.
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Health in Women | At the baseline.
  SF-36v Health Survey developed by RAND Corporation measures Functional Health form. The measure the participants' perspective. The 36 item questionnaire developed by the Rand Corporation taps eight health concepts including physical well being; bodily pain; role limitations;emotional problems; energy/ fatigue; general health perceptions. Each item is scored on a Likert scale o 1-4 with a higher score indicative of higher functional health with the possible score range from 36-144.
Power to change in Women | At the baseline.The tool is nown as the Power as Knowing Participation in Change Tool (PKPCT).
  Power as Knowing Participation in Change (PKPCT this measure measures power defined as the capacity to participate knowingly in the nature of change as manifest by awareness of choices, freedom to act intentionally and involvement in creating change. this is a seven point semantic differential scale consisting of 12 bipolar adjective pairs and one repeat adjective pairas a retest. The score range is 12 to 84 lower score indicates lower power higher score indicates higher power.
Functional Health in Women | Twenty-one days after the baseline, change will be measured over time
  SF-36v, Health Survey-Functional Health from the Participants' Perspective
Power to Change in Women | Twenty-one days after the baseline, change will be measured over time
  Power as Knowing Participation to change (PKPCT)

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis S Hansell, Principal Investigator — Seton Hall University
Locations (2):
- United States (2):
  - Seton Hall University, College of Nursing, Nutley, New Jersey
  - Seton Hall University, IHS Campus, Nutley, New Jersey

IPD SHARING:
Plan to Share IPD: No
Data will not be shared and be held in strict confidentiality.

REFERENCES:
- [Background] Barrett EA. Power as knowing participation in change: what's new and what's next. Nurs Sci Q. 2010 Jan;23(1):47-54. doi: 10.1177/0894318409353797. PMID 20026728
- [Background] Caroselli C, Barrett EA. A review of the power as knowing participation in change literature. Nurs Sci Q. 1998 Spring;11(1):9-16. doi: 10.1177/089431849801100105. PMID 9555424
- [Background] Hansell PS, Hughes CB, Caliandro G, Russo P, Budin WC, Hartman B, Hernandez OC. The effect of a social support boosting intervention on stress, coping, and social support in caregivers of children with HIV/AIDS. Nurs Res. 1998 Mar-Apr;47(2):79-86. doi: 10.1097/00006199-199803000-00006. PMID 9536191
- [Background] Malicki J. The accuracy of dose determination during total body irradiation. Strahlenther Onkol. 1999 May;175(5):208-12. doi: 10.1007/BF02742397. PMID 10356609
- [Background] Giacobbi PR Jr, Stewart J, Chaffee K, Jaeschke AM, Stabler M, Kelley GA. A Scoping Review of Health Outcomes Examined in Randomized Controlled Trials Using Guided Imagery. Prog Prev Med (N Y). 2017 Dec;2(7):e0010. doi: 10.1097/pp9.0000000000000010. PMID 29457147
- [Background] Hong, S.H. (2013) The relationship between perceived health status and health promoting behaviors among nursing students. Journal of Korean Academy Society in Nursing Education 19, 78-86.
- [Background] Park, S.; Lee, Y.H. (2016) Effects of perceived health status, health attitude, and health concern on health promoting behavior in adults. Journal of Korea Contents Association, 16, 192-202.
- [Background] Pender, N.J.; Murdaugh, C.L.; Parsons, M.A. (2010) Health Promotion in Nursing Practice, 6ᵗʰ edition; Prentice-Hall: Upper Saddle River, N.J.
- [Background] Zech N, Hansen E, Bernardy K, Hauser W. Efficacy, acceptability and safety of guided imagery/hypnosis in fibromyalgia - A systematic review and meta-analysis of randomized controlled trials. Eur J Pain. 2017 Feb;21(2):217-227. doi: 10.1002/ejp.933. Epub 2016 Nov 29. PMID 27896907